CLINICAL TRIAL: NCT06589115
Title: Blood Flow Restriction Therapy Improves Tibial Plateau Fracture Recovery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn prior to enrollment due to lack of available financial resources.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Elizabeth Nolte, Principal Investigator, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00047532
Record Dates: First submitted 2024-07-15; First posted 2024-09-19 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Tibial Plateau Fractures
MeSH Terms: conditions — Tibial Plateau Fractures | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation Protocol (Active Comparator): Standard physical therapy will be performed according to the clinic standard with manual lymphatic drainage, cryotherapy, and 20 minutes of physical therapy two times a week for fourteen weeks following the initial post-operative visit.
  Interventions: Other: Physical Therapy
- Rehabilitation Protocol and Blood Flow Restriction (Experimental): In addition to the standard physical therapy, the blood flow restriction group will also begin standard physical therapy care supplemented with blood flow restriction therapy two times a week for 10 weeks after wound healing.
  Interventions: Other: Blood Flow Restriction Cuff; Other: Physical Therapy

INTERVENTIONS:
Other: Blood Flow Restriction Cuff — The standardized exercises will be performed while wearing a blood flow restriction cuff.
  Arms: Rehabilitation Protocol and Blood Flow Restriction
Other: Physical Therapy — Standard physical therapy

SUMMARY:
The goal of this clinical trial is to investigates the effectiveness of physical therapy augmented with blood flow restriction (BFR) therapy relative to standard physical therapy in patients after an open reduction and internal fixation of a closed tibial plateau fracture.

The main aims are:

* Collect functional and patient self-reported outcomes data
* Assess leg muscle atrophy
* Acquire motion analysis dynamics and knee strength data.

Participants will be randomized into either a rehabilitation protocol or that protocol with blood flow restriction and be followed for 1 year.

DETAILED DESCRIPTION:
Standardized Surveys: Participants will complete two patient reported functional outcome assessments via questionnaires, the KOOS (Knee Injury and Osteoarthritis Outcome Score) and the PROMIS PF (Patient-Reported Outcomes Measurement Information System Physical Function). The PROMIS PF is a computer adaptive, reliable, and validated instrument used to evaluate patient-reported outcome measures regarding physical function ranging from low to very high, along with mental and social well-being. The KOOS is a knee-specific self-administered questionnaire that assesses five long-term and short-term outcomes of knee injury: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life.

Blood Flow Restriction Cuff: Along with standard physical therapy, three of the standardized exercises will be performed while wearing an Owens Delfi blood flow restriction cuff (Delfi Medical, San Antonio, TX). To attain partial vascular occlusion, an easy-fit nylon cuff (11.5 cm x 86 cm, 5mm thick) will be placed as proximal as possible on the patient's thigh of the involved leg. Total limb occlusion pressure will be individualized and set between 60% to 80% of the complete arterial occlusion pressure. Limb occlusive pressure will be calculated with the participants in the position for exercise to ensure accurate calculation of limb occlusive pressure. This individual approach prevents excessive pressure in individuals with lower limb occlusion pressures.

Tape Measure: A non-elastic, flexible plastic tape measure will be used. The thigh circumference will be measured at a point 15 cm proximal to the superior pole of the patella. Calf circumference will be measured at the point of greatest circumference while subjects are supine with the knee extended; subcutaneous tissues will not be compressed.

Motion Analysis: Quantitative motion analysis will be conducted at the Medical College of Wisconsin (MCW) Center for Motion Analysis (CMA) using a motion analysis camera system and wireless surface electromyography (EMG) electrodes to determine temporal-spatial parameters, kinematics, kinetics, and muscle activity during walking, sit-to-stand, forward lunge, and step-up-and-over tasks. A validated standardized gait model will be used.

Leg Strength Assessment: Isometric, concentric and eccentric strength will be assessed using the Biodex System 3 Pro dynamometer. Each subject will undergo bilateral leg strength testing.

ELIGIBILITY:
Inclusion Criteria:

1. Equal to or greater than 18 years of age
2. ORIF (open reduction and internal fixation) of a closed unicondylar tibial plateau fracture
3. Planning to attend physical therapy at one of the eligible Froedtert locations with BFR therapy capabilities

Exclusion Criteria:

1. Patient is unable to provide consent
2. At time of tibial plateau fracture has evidence of a(n)

   1. Open fracture(s)
   2. Fracture(s) with associated vascular injury,
   3. Fracture(s) with extensive soft tissue injury preventing the ability to apply a tourniquet
   4. Ipsilateral or contralateral lower extremity fracture(s)
   5. Pelvic or spinal trauma
3. History of deep venous thrombosis (DVT)
4. History of peripheral vascular disease
5. Body Mass Index > 40
6. Any history of condition that would affect the patient's ability to bear weight as tolerated post-operatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Collect participant knee injury consequences questionnaire | Prior to initiation of therapy, and 3, 6, and 12 months postoperatively
  Participants will complete the KOOS (Knee Injury and Osteoarthritis Outcome Score) questionnaire.
Collect participant reported function outcome questionnaire | Prior to initiation of therapy, and 3, 6, and 12 months postoperatively
  Participants will complete the PROMIS PF (Patient-Reported Outcomes Measurement Information System Physical Function) questionnaire.
Assess leg muscle atrophy | Prior to initiation of therapy and 3, 6, and 12 months postoperatively
  Bilateral thigh and calf circumferential girth measurements will be taken once prior to initiation of therapy and then additionally at 3, 6, and 12 months postoperatively as a surrogate for muscle mass.
Acquire motion analysis dynamics | 6 and 12 months postoperatively.
  Participants will undergo 3D motion analysis with concurrent surface EMG (i.e., the electrical activity of the muscle) during walking, sit-to-stand, forward lunge, and step-up-and-over tasks.
Acquire knee strength data. | 6 and 12 months postoperatively.
  Bilateral knee strength (i.e., muscle force production) will be assessed for isometric, concentric and eccentric muscle contractions using a Biodex dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Nolte, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States